CLINICAL TRIAL: NCT05866653
Title: Effect of Lidocaine Transdermal Patch as Add-On Therapy in Treatment of Oxaliplatin Induced Peripheral Neuropathy in Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sharmeen Tania Shovah, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BSMMU/20023/265
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Oxaliplatin Induced Peripheral Neuropathy in Cancer Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Active Comparator): This group will consist of 45 patients who are scheduled to receive oxaliplatin based chemotherapy regimen. After receiving 2 cycles of chemotherapy usually patient develops OIPN. Patients who will develop OIPN with pain intensity ≥4 in VAS scores will be included. The patients will be treated with one lidocaine transdermal patch/day for 12 hours for 10 days as add on therapy with standard treatment by oncologist.
  Interventions: Drug: lidocaine transdermal patch
- Placebo Arm (Placebo Comparator): This group will consist of 45 patients who are scheduled to receive oxaliplatin based chemotherapy regimen. After receiving 2 cycles of chemotherapy usually patient develops OIPN. Patients who will develop OIPN with pain intensity ≥4 in VAS score will be included. The patients will be treated with one placebo patch/day for 12 hours for 10 days as add on therapy with standard treatment by oncologist.
  Interventions: Drug: lidocaine transdermal patch

INTERVENTIONS:
Drug: lidocaine transdermal patch — The topical pain-relieving treatment 5% lidocaine transdermal patch has been registered in the USA since 1999

SUMMARY:
Oxaliplatin (OXA) is a third-generation platinum-based chemotherapeutic drug with better efficacy for colorectal carcinoma (CRC). Oxaliplatin-induced peripheral neuropathy (OIPN) is one of the most frequent dose-limiting or even treatment-terminating side effects that impair optimal treatment regimens in a significant proportion of patients from 19% to over 85%. Thus, OIPN impacts the quality of life and the patient's survival. OIPN is a clinical challenge and healthcare professionals are facing this challenge with a limited selection of analgesics and nonpharmacological therapies. Pregabalin is a structural derivative of GABA and is one of the effective treatment modalities for OIPN. It binds with high affinity to the alpha2-delta site of voltage-gated calcium channels in central nervous system tissues and inhibits neurotransmitter release, thus producing anti-nociceptive and anti-seizure effects.

DETAILED DESCRIPTION:
Oxaliplatin (OXA) is a third-generation platinum-based chemotherapeutic drug with better efficacy for colorectal carcinoma (CRC). Oxaliplatin-induced peripheral neuropathy (OIPN) is one of the most frequent dose-limiting or even treatment-terminating side effects that impair optimal treatment regimens in a significant proportion of patients from 19% to over 85%. Thus, OIPN impacts the quality of life and the patient's survival. OIPN is a clinical challenge and healthcare professionals are facing this challenge with a limited selection of analgesics and nonpharmacological therapies. Pregabalin is a structural derivative of GABA and is one of the effective treatment modalities for OIPN. It binds with high affinity to the alpha2-delta site of voltage-gated calcium channels in central nervous system tissues and inhibits neurotransmitter release, thus producing anti-nociceptive and anti-seizure effects. But it has dose related side effects and intolerability Clinical data shows that administration of pregabalin tablet 150mg/day for 2-6 weeks significantly improves the neuropathy induced by oxaliplatin in 48% of the patients. Lidocaine transdermal patch (L5%P) is a local anesthetic medication with analgesic effect. It works in a different mechanism from pregabalin by stopping nerves from sending pain signal by blocking sodium ion channel, thus reduces ectopic nerve discharges, relieves hyperalgesia and modulates the inflammatory response. It is applied on most painful area on skin and shows further benefits as low systemic absorption (3-5%), reduced risk of systemic toxicity, minimized side effects and reduced potential of drug interactions. Clinical data have indicated its efficacy in neuropathic pain conditions (PHN), including diabetic polyneuropathy (DPN) and herpes zoster neuralgia. Moreover, Lidocaine inhibits proliferation and induces apoptosis in colorectal cancer cells by up regulating mir-520a-3p and targeting EGFR. No study has been conducted yet to determine the effect of lidocaine patch on OIPN but theoretically it might be a potentially useful treatment option. This proposed study is therefore an effort whether there is any role of lidocaine patch in symptomatic improvements of OIPN as add on therapy with pregabalin tablet. This study will be a randomized, double-blind, placebo controlled clinical trial. It will be conducted in the department of pharmacology, BSMMU in collaboration with National institute of cancer research and hospital (NICRH) from the day of approval by the IRB to July, 2023. A total of ninety (90) patients from indoor department of clinical oncology will be selected for the study according to inclusion and exclusion criteria. After receiving oxaliplatin treatment regimen and after development of OIPN with pain intensity ≥ 4 in VAS scores at baseline, participants will randomly be assigned into two intervention groups. Group A (45) will receive lidocaine transdermal patch (1 patch/day for 12 hours) along with pregabalin tablet (75mg/day) for 10 days and group B (45) will receive placebo patch (1patch/day for12 hours) along with pregabalin tablet (75mg/day) for 10 days. Every cycle interval consists 3 weeks and assessment of OIPN will be done at baseline and after 3rd and 6th weeks. Quality of life will be measured by FACT/GOG-NTX neurotoxicity scoring and severity of neuropathy by NCI-CTCAE grading scale. Comparison between the effects of interventions in two groups can be made by using data collected from each group

ELIGIBILITY:
Inclusion Criteria:

* Adults with stage II, III and IV colorectal cancers, scheduled to receive an oxaliplatin-based chemotherapy regimen.
* Patients could be receiving concomitant chemotherapy.
* Patient ECOG performance status 0-3.

Exclusion Criteria:

* • Pre-existing symmetric peripheral painful neuropathy due to diabetes mellitus or other causes.

  * Presence of brain metastases.
  * Renal insufficiency (calculated creatinine clearance<30ml/min).
  * Moderate to severe hepatic insufficiency (ALTor AST >3times upper level of normal if no liver metastases are present; ALTor AST >5 times upper limit of normal if liver metastases are present).
  * Current uncontrolled cardiac arrhythmias (non-sinus rhythm).
  * Any topical treatment with other medication for neuropathic pain.
  * Pregnancy or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Visual Analogue Scale (VAS) pain score | From the baseline assessment to 3 and 6 weeks
  Measure pain

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code